CLINICAL TRIAL: NCT02899832
Title: A Study of Hemodynamic Changes Using Near Infra-red Spectrometry (NIRS) in Infantile Epilepsy Spasms
Acronym: SPASMES-NIRS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2012_843_0029
Record Dates: First submitted 2016-09-05; First posted 2016-09-14 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Epilepsy
Keywords: children; spasms
MeSH Terms: conditions — Epilepsy; Spasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- NIRS: Near Infra Red Spectroscopy.
  Interventions: Device: NIRS

INTERVENTIONS:
Device: NIRS — Near Infra Red Spectroscopy

SUMMARY:
This study will included 20 children presenting with epilepsy with spasms. It aims to offer these children, non invasively and without supplementary examinations, a recording of local and cerebral hemodynamic changes concomitant with an electroencephalographic recording during epileptic episodes. This will be carried out by combining optical imaging using near infra-red spectroscopy (NIRS) with electroencephalography (EEG), in a simultaneous high-resolution (HR) recording.

This study is among those based on multimodal analyses of epilepsy, combining methods of analysis of electrical activity (electrical imaging) and hemodynamics (optical imaging).

Surface electroencephalography (EEG) is a precious tool enabling the study of neuronal dysfunction from a functional point view. It is used in the routine follow-up of children with epilepsy. Optical imaging is a promising medical imaging technique. It uses light in the spectral regions of near infra-red as a source of radiation. It is quantitative, rapid, non invasive, and inoffensive which could easily be used at the child's bedside or in a clinical setting and can provide metabolic information about cerebral function.

This study is multidisciplinary, which calls upon the skills of neurophysiologists, biophysicists, and clinicians

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 and 6 years old presenting infantile spasms according to the Classification of the International League Against Epilepsy

Exclusion Criteria:

* Children younger than 3 months and older than 6 years of age, refusal of one of the parents, and dermatosis of the scalp

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between 3 and 6 years old presenting infantile spasms
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-02-21 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
changes in HbO | Day 0
  hemodynamic changes in [HbO] before spasms, during spasms, and after spasms
changes in Hbr | Day 0
  hemodynamic changes in [Hbr] before spasms, during spasms, and after spasms

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice WALLOIS, MD, PhD, Principal Investigator — CHU Amiens
Locations (2):
- France (2):
  - CHU Amiens, Amiens
  - Fondation Ophtalmologique Rothshild, Paris